CLINICAL TRIAL: NCT04615260
Title: Comparison of Fusion Success Between NanoBone Synthetic Bone Graft and Local Autogenous Bone Graft in Posterolateral Spinal Fusion
Brief Title: Rate of Bony Fusion Using NanoBone® Synthetic Bone Graft Versus Local Autologous Bone Graft.
Acronym: BONE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artoss Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H0015310
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis
Keywords: Nanotechnology; NanoBone; Spine Fusion; Bone Graft
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: Study is a prospective, non-randomized, single center clinical investigation. Each subject will serve as their own control during this study, as patients will receive the Nanobone graft on the right side of their spine and the local bone graft on their left side.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm subject is own control (Other): Posterolateral fusion is bilateral, patients will receive the Nanobone graft on the right side of their spine and the local bone graft on their left side.
  Interventions: Device: NanoBone

INTERVENTIONS:
Device: NanoBone — Nanobone® Synthetic Bone Graft is a nanocrystalline hydroxyapatite imbedded in a silica gel matrix. The nanocrystalline structure accurately replicates autologous hydroxyapatite and the silica gel matrix that rapidly transforms into an osteogenic matrix post-implantation. NanoBone promotes remodeling by acting as a strong osteoinductive material. NanoBone® is available as a putty.
  Other Names: NanoHA (SiO2)

SUMMARY:
The objectives of this longitudinal study are to assess and measure fusion status (fused or not fused) and rate of bony fusion using NanoBone® Synthetic Bone Graft in patients requiring one to two level lumbar posterolateral fusion procedures with or without commercially available rigid spinal instrumentation. Our hypothesis is that the Nanobone synthetic bone graft will be as effective at creating a fusion in the lumbar spine as compared with a local bone graft. Each subject will serve as their own control during this study, as patients will receive the Nanobone graft on the right side of their spine and the local bone graft on their left side.

DETAILED DESCRIPTION:
Subjects will be recruited for this study from among those scheduled to undergo 1-2 level posterolateral spinal fusion procedures with bone grafting for degenerative disc disease or grade 1-3 spondylolisthesis. The study will entail each subject having a local bone graft placed on the left side of their spine, with Nanobone placed on the right side of their spine during the procedure. Eligible and consenting patients recruited for this study will be subject to the standard of care. This includes the following visits: preoperative, operative, post-discharge, 4 months postoperative, 1-year postoperative, and 2-years postoperative. They will be subject to standard of care imaging modalities including AP, lateral, and flexion/extension lumbar radiographs at pre-operative, post-discharge, 4-months postoperative, 1-year postoperative, and 2-year postoperative time points. Standard of care advanced imaging including a CT scan or magnetic resonance imaging (MRI) scan will be performed pre-operatively. Patients will also receive standard of care clinical examinations and self-assessments at all clinic visits. Imaging obtained outside the standard of care for this study will include 1-year and 2-year lumbar CT scans to evaluate fusion. The 2-year lumbar CT scan will only be required if fusion has not been demonstrated at the time of the 1-year lumbar CT scan. Patients enrolled in this study who are treated with rigid pedicle screw fixation must be treated using rigid pedicle screw instrumentation appropriate for posterolateral spinal fusions.

ELIGIBILITY:
Inclusion Criteria:

1. The individual has signed and dated a study specific informed consent form approved by the Institutional Review Board at UMMHC.
2. The individual is 18 to 85 years of age.
3. The individual is skeletally mature.
4. The individual has been diagnosed with 1 or 2 level degenerative disc disease or spondylolisthesis grade 1-3 with or without spinal stenosis, requiring posterolateral spinal fusion surgery with bone grafting.
5. The individual is physically and mentally willing and able to comply with the postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. The individual has had any previous attempts at fusion, at any lumbar levels.
2. The individual is morbidly obese (defined as 100 lbs over the recommended ideal weight as described in the Metropolitan Life Height and Weight Tables for Men and Women and or having a BMI >39).
3. Patients with osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated.
4. Patients with systemic collagen, bone or mineralization dysfunction (such as Paget's disease, osteogenesis imperfecta, Ehlers-Danlos Syndrome).
5. Patients who suffer from uncontrolled diabetes mellitus type I or insulin-dependent diabetes mellitus type II. (definition based on the glycosylated Haemoglobin level)
6. Patients who are suffering from autoimmune disease.
7. Patients who previously underwent chemotherapy, immunosuppressive disease or radiation to the local area.
8. Patients who received or are currently receiving corticosteroids (> 2 years > 5 mg prednisolone equivalent/d).
9. Patients with active local or systemic infection.
10. Patients with any known active malignancy.
11. Patients with other concurrent physical or mental conditions which are likely to affect their outcome.
12. Patient unable to consent for themselves
13. Pregnant women
14. Non-English speaking subjects. These subjects are excluded because they would not be able to complete the English-language surveys required during this study. Only English language versions of these surveys have been validated.
15. Prisoners
16. Patients less than 18 years old

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion | 12 months
  Fusion will be defined as:
  * Evidence of bridging trabecular bone between the transverse processes of the involved vertebral bodies
  * Translational motion < 3.5mm on flexion/extension radiographs; and
  * Angular motion <5 degrees on flexion/extension radiographs.
Oswestry Disability Index (ODI) 0% lowest, no disability to 100% disabled, bedridden | 12 months
  Change from pre-operative score

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) 0-no pain to 10-worst possible pain | 12 months
  Change from pre-operative score
SF-36 (Short Form 36) | 12 months
  Change from pre-operative score

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Connelly, MD, Principal Investigator — UMass Memorial Health
Locations (1):
- UMass Memorial Health Care, Worcester, Massachusetts, United States